CLINICAL TRIAL: NCT01112371
Title: A Prospective, Single-center, Randomized, Parallel Group Trial to Investigate the Efficacy of Contractubex® Gel, Containing Extractum Cepae, Allantoin, and Heparin, in Scars After Abdominal Caesarean Section
Brief Title: Contractubex Treatment in Scars After Abdominal Caesarean Section
Acronym: ConMex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 90011_4023_1
Record Dates: First submitted 2010-04-06; First posted 2010-04-28 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Scars
Keywords: scars after abdominal Caesarean section
MeSH Terms: conditions — Cicatrix | interventions — allantoin, heparin, onion extract drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contractubex (Experimental)
  Interventions: Drug: Contractubex
- Non treatment (No Intervention)

INTERVENTIONS:
Drug: Contractubex — Contractubex® Gel, containing 10% extractum cepae, 1% allantoin and 50/U of sodium heparin per one gram of gel.
  Active drug group: The gel will be applied twice daily (morning/evening). Approximately 2 cm of the IMP are applied onto the scar by light massage rubbing carefully until the product is worked in.
  Other Names: Other names have not been specified.
  Arms: Contractubex

SUMMARY:
The purpose of this study is to investigate the efficacy of Contractubex® Gel, containing extractum cepae, allantoin and heparin, in the treatment of scars after abdominal Caesarean section compared to untreated scars after abdominal Caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Females having given birth via elective abdominal Caesarean section for the first time within the last 5 to 10 days who had their suture removed (removed at screening).
* Age: 18 years or older.
* The subject must be willing and must be able to complete the entire course of the trial and to comply with the trial instructions.
* Written informed consent has been obtained from the subject.
* Females using suitable contraceptions.

Exclusion Criteria:

* Use of any inadmissible medication, e.g. systemic corticosteroids, systemic immunosuppressants (such as cytostatics, therapy with antibodies, biologics, interferone, mykophenolatmofetil, methotrexate, cyclosporine, azathioprine). Any additional topical treatment in the area of the lower abdomen, regardless of the mode of action.
* Any other planned topical treatment in the lower part of the abdomen during the course of the trial.
* Any infection or wound in the area to treat.
* History of keloids or hypertrophic scars.
* Any severe or uncontrolled systemic disease (e.g. cardiac, renal, pulmonary, hepatic, or gastrointestinal), malignant tumor, or medical history of HIV infection.
* Any tumor diseases in the abdominal region independent of their dignity.
* Females having given birth via emergency abdominal Caesarean section.
* Psychiatric problems which, in the investigator's opinion, are severe enough to interfere with the trial results.
* Participation in another clinical trial within 30 days prior to screening.
* Evidence or suspicion that the subject might not comply with the study directives and/or that she is not reliable or trustworthy.
* Evidence or suspicion that the subject is not willing or unable to understand the information given to her as part of the informed consent, in particular regarding the risks and discomfort to which she would agree to be exposed.
* Previous participation in this clinical study.
* Known allergy or hypersensitivity to the study drug(s) or one of the ingredients of the formulation.
* Subjects who are imprisoned or are lawfully kept in an institution.
* Employees or direct relatives of an employee of the CRO, the study center or Merz Pharmaceuticals.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Appearance of the scars will be evaluated by use of the Patient and Observer Scar Assessment Scale [POSAS]. | Screening and 12 weeks
  The scale consists of two numeric scales which need to be filled out by the observer and the patient, respectively.

SECONDARY OUTCOMES:
Appearance of the scars will be evaluated by use of the Patient and Observer Scar Assessment Scale [POSAS]. | Screening and 6 weeks
  The scale consists of two numeric scales which need to be filled out by the observer and the patient, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Ocampo Candiani, MD, Principal Investigator — Jefe del Departamento Dermatologia, Facultad de medicina y Hospital Universitario, Universidad Autonoma de Nuevo León, Monterrey Nuevo León,C.P. 64460, Mexico
Locations (1):
- Jefe del Departamento Dermatologia, Facultad de medicina y Hospital Universitario, Universidad Autonoma de Nuevo León, Monterrey Nuevo León, C.p., Mexico

REFERENCES:
- [Result] Ocampo-Candiani J, et al. Efficacy of a topical gel containing extractum cepae, allantoin and heparin in the treatment of abdominal caesarean section scars. IMCAS Annual Meeting 2013. www.imcas.com/en/imcas2013/schedule/lecture/id/5971
- [Result] Ocampo-Candiani J, Vazquez-Martinez OT, Iglesias Benavides JL, Buske K, Lehn A, Acker C. The prophylactic use of a topical scar gel containing extract of Allium cepae, allantoin, and heparin improves symptoms and appearance of cesarean-section scars compared with untreated scars. J Drugs Dermatol. 2014 Feb;13(2):176-82. PMID 24509969